CLINICAL TRIAL: NCT01285583
Title: An Open-label Safety Extension Study of TRO19622 in Amyotrophic Lateral Sclerosis (ALS) Patients Treated With Riluzole
Brief Title: Safety Extension Study of TRO19622 in ALS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: WN29852; TRO19622 CL E Q 1425-1 (Other: trophos id)
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophoc Lateral Sclerosis; TRO19622; Olesoxime; Trophos
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — olesoxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olesoxime (Other): All patients will receive the IMP as add-on to riluzole 50 mg bid orally, 50 mg morning and evening on an empty stomach ie at least 20 min before the meal.
  Interventions: Drug: TRO19622

INTERVENTIONS:
Drug: TRO19622 — 2 capsules of TRO19622 (330mg) once a day with the noon meal as add-on therapy to riluzol 50mg bid

SUMMARY:
The purpose of the assay is to assess the safety of TRO19622 330 mg QD as add-on therapy to riluzole 50 mg bid in the treatment of patients suffering from ALS, after completion of the preceding clinical trial (TRO19622 CL E Q 1015-1) in an open label extension.

DETAILED DESCRIPTION:
Entry of a patient into this safety study is intended to occur immediately after the patient has finished participating in the preceding efficacy study (Protocol TRO19622 CL E Q 1015-1).

The Investigator will explain to the patients the nature of this open-label safety study, its procedures, requirements and restrictions so as to obtain their written informed consent.

Each patient will be treated with olesoxime (TRO19622) until the results of the double-blind trial become available with a maximum of 15 months.

Follow-up visits will take place every 3 months (+/- 2 weeks).

Safety assessments will be performed at all visits (every 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the 18-month safety and efficacy study of TRO19622 in Amyotrophic Lateral Sclerosis (ALS) patients treated with riluzole (Protocol TRO19622 CL E Q 1015-1).
* Both the investigator and the patient will decide based on previous good tolerance and other clinical grounds whether or not to participate to the open-label extension.
* If patients were on anti-vitamin K during the double-blind period, when entering the open-label extension, coagulation tests should be monitored in exactly the same conditions as if a new anticoagulant treatment was initiated and the dose of anti-vitamin K should be adjusted accordingly.
* Patients enrolling from this prior safety and efficacy study must:

  * If female of childbearing age of potential, continue to use adequate birth control methods and have a negative serum pregnancy test at the preceding double-blind protocol termination visit. Male and female partners must agree to use an effective method of birth control during their participation in the trial and for at least 15 days after the last IMP dose. Both partners must use reliable methods of contraception with 2 independent methods. The following measures are acceptable: Hormone contraceptives (e.g. oral contraceptives or comparable methods), intrauterine device, condoms with spermicidal coating or in combination with spermicidal creams, total abstinence or sterilisation performed in the past.
  * Be able to follow the investigator's instructions and be able to comply with the visit schedule and visit requirements; and
  * Sign a written informed consent.

Exclusion Criteria:

Patients may not participate in this study if they have an ongoing, unresolved, clinically significant medical problem (including patients having experienced serious adverse events or non-serious, but medically significant adverse events during the preceding safety and efficacy study that was assessed to be related to the study medication by the investigator) that in the judgment of the investigator would make it unsafe for the patient to participate in the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the safety assessment. | Safety assessment will be calculated from the date of enrollment for a maximum of 15 months.
  safety criteria will be:
  * Occurrence of AEs,
  * Physical examination,
  * Laboratory tests,
  * Vital signs and ECG,

SECONDARY OUTCOMES:
Secondary Outcome Measures | Every 3 month, from the date of enrollment for a maximum of 15 months.
  Secondary Outcome Measures will be:
  * Survival time
  * Total score of the 48-point ALS Functional Rating Scale Revised
  * Slow Vital capacity (SVC) as a percentage of predicted SVC only if the SVC is performed by the site in a routine-way during standard ALS visit. This test will not be performed for the sole purpose of the study

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Meininger, MD, PhD, Principal Investigator — Groupe Hospitalier Pitie-Salpetriere
Locations (15):
- University Hospital Gasthuisberg - Dept Neurology - Herestraat 49, Leuven, Belgium
- France (7):
  - HCL Hôpital Neurologique et Neurochirurgical Pierre Wertheimer - Neurologie C et Laboratoire d'électromyographie - 59, boulevard Pinel, Bron
  - CHRU de LILLE - Hôpital Roger Salengro - Centre SLA-MMN - Sce de Neurologie et Pathologie du Mouvement, Lille
  - Centre SLA Limoges - Service de Neurologie, Limoges
  - Hôpital La Timone - Service Neurologie et Maladies Neuromusculaires, Marseille
  - Clinique du Motoneurone - Sce d'Explorations Neurologiques - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nice - Hôpital de l'Archet 1 - Centre de Référence pour les Maladies Neuromusculaires et la SLA, Nice
  - Groupe Hospitalier PITIE-SALPETRIERE - Fédération des Maladies du Système Nerveux, Paris
- Germany (4):
  - Charité Universitätsmedizin Berlin, Campus Virchow-Klinikum, Neurologische Poliklinik Ambulanz für ALS und andere Motoeneuronenerkrankungen, Berlin
  - Universitätsklinik und Poliklinik für Neurologie - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Neurologische Klinik Medizinische Hochschule, Hanover
  - Universitäts- und Rehabilitationskliniken Ulm (RKU) - Neurologische Universitätsklinik, Ulm
- Hospital Carlos III - Unidad de ELA - Sinesio Delgado, 10, Madrid, Spain
- United Kingdom (2):
  - King's MND Care and Research Center - Academic Neurosciences Building PO Box 41 Institute of Psychiatry, London
  - Academic Neurology Unit - University of Sheffield - Section of Neuroscience - Division of Genomic Medicine - School of Medicine and Biomedical Sciences, Sheffield